CLINICAL TRIAL: NCT01217424
Title: Is Reflexology as Effective as Aromatherapy Massage for Symptom Relief in an Outpatient Oncology Population?
Brief Title: Reflexology or Aromatherapy Massage in Relieving Symptoms in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000686459; RMNHS-REFLEXOLOGY; EU-21075; MREC-10/H0801/31
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Pain; Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; pain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Pain | interventions — Aromatherapy; Massage; Psychiatric Rehabilitation; Musculoskeletal Manipulations

INTERVENTIONS:
Other: questionnaire administration
Procedure: aromatherapy and essential oils
Procedure: management of therapy complications
Procedure: massage therapy
Procedure: psychosocial assessment and care
Procedure: reflexology procedure

SUMMARY:
RATIONALE: Reflexology and aromatherapy massage may lessen symptoms in patients with cancer. It is not yet known whether reflexology is more effective than aromatherapy massage in relieving symptoms in patients with cancer.

PURPOSE: This randomized clinical trial is studying reflexology to see how well it works compared with aromatherapy massage in relieving symptoms in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether reflexology is as effective as aromatherapy massage for alleviation of self-selected symptoms in patients with cancer in an outpatient setting.

Secondary

* To determine the difference between the two therapies with respect to Visual Analogue Scale (VAS) relaxation scores before and after each treatment.

OUTLINE: Patients are stratified according to gender (male vs female), treatment (chemotherapy vs other) and their first concern choice (pain vs other). Patients are randomized to 1 of 2 intervention arms.

* Arm I (Reflexology): Patients undergo 45-60 minutes of reflexology for 4 sessions.
* Arm II (Aromatherapy massage): Patients undergo 45-60 minutes of of aromatherapy massage for 4 sessions.

Patients complete questionnaires (Measure Yourself Concerns and Well-being [MYCAW] questionnaire and Visual Analogue Scale [VAS]) at baseline, before and after each session, and after completion of all four sessions.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Any patient receiving treatment for cancer at the Royal Marsden NHS Foundation Trust Hospital

  * Must be attending the hospital as an outpatient
* Planning to access complementary therapy

PATIENT CHARACTERISTICS:

* No excessive pain in both hands and both feet
* Not experiencing a combination of conditions affecting both hands and both feet which would prevent reflexology of either hands or feet from taking place, including any of the following:

  * Deep vein thrombosis
  * Lymphedema
  * Infected or broken skin
  * Recent scars or injuries
  * Phlebitis
  * Areas currently receiving radiotherapy (or received radiotherapy in the past 2 weeks)
* Able and willing to attend the hospital for four 1-hour sessions

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 months since prior and no other concurrent massage therapy or reflexology at the Royal Marsden NHS Foundation Trust Hospital or from another practitioner
* Not planning to undergo massage therapy or reflexology while also taking part in this study
* At least 2 months since prior and no other concurrent massage therapy at the Royal Marsden NHS Foundation Trust Hospital

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Difference of 1 point of concern scores in Measure Yourself Concerns and Well-being (MYCAW) questionnaire from baseline to second evaluation (after completion of all four sessions of therapy)

SECONDARY OUTCOMES:
Difference of 2 points of concern scores in MYCAW questionnaire
Difference in MYCAW overall well-being score
Change over time in pre-session Visual Analogue Scale (VAS) relaxation score (long-term relaxation benefit)
Change in pre- to post-session VAS relaxation score (short-term relaxation benefit)
Percentage of patients gaining benefit from the intervention defined as improvement by at least 1 point in all answered MYCAW scales

CONTACTS AND LOCATIONS:
Overall Officials: Clare Shaw, MD, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - London, London, England, United Kingdom